CLINICAL TRIAL: NCT06803459
Title: Effects of Baduanjin and Proprioceptive Neuromuscular Facilitation on Upper Crossed Syndrome Among University Students in Henan Province，China
Brief Title: Effects of Baduanjin and PNF on Upper Crossed Syndrome Among University Students in Henan Province，China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Long Canghao, students, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20230067
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-10

CONDITIONS: Upper Crossed Syndorme
Keywords: UCS

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Baduanjin (Experimental): This will be an experiment of about 60 minutes three times a week for 12 weeks.
  Interventions: Other: Baduanjin; Other: PNF
- PNF (Experimental): This will be an experiment of about 60 minutes three times a week for 12 weeks.
  Interventions: Other: Baduanjin; Other: PNF
- Control Group (No Intervention): The subjects performed daily activities for 12 weeks.

INTERVENTIONS:
Other: Baduanjin — 36 times.
  Arms: Baduanjin; PNF
Other: PNF — 36 times.
  Arms: Baduanjin; PNF

SUMMARY:
Upper crossed syndrome (UCS) is a condition threatening the physical health, anxiety level and quality of life of university students. Despite biomechanical and neurological approaches are available, evidence on their practicality and effectiveness remained scarce among university students. This randomized controlled trial aimed to determine the effectiveness of Baduanjin and Proprioceptive neuromuscular facilitation (PNF) on symptoms of UCS in university students in Henan Province, China. A total of 90 university students with crossed syndrome will be recruited and randomised into intervention (Baduanjin and PNF) and control groups. The intervention groups will undergo a structured exercise therapy or PNF for 12 weeks. The primary outcomes are improvement on neck range of motion and static posture while secondary outcomes are perceived Quality of Life (QoL) and level of anxiety.

DETAILED DESCRIPTION:
In this study, the comparative design is referred to as a descriptive approach because of its appropriateness. This study was conducted primarily through an experimental intervention. It was a randomized controlled trial of 12 weeks duration. In this process, the research instruments and markers were prepared and then during the experiment, the comparative study was a descriptive comparative method, which was mainly described by comparing the changes in data before and after the experiment. This study includes three main aspects of the variable study. The first aspect was the range of motion of the neck joints, which consisted of six main variables: head extension, posterior extension, left extension, right extension, left rotation, and right rotation. The second aspect is the static postural index of patients with upper crossed syndrome. The FHA and FSA variables were selected for assessment in this study. The third aspect is the rating of patients' self-perceptions before and after the experiment, including the degree of cervical pain, the degree of cervical disability and the degree of anxiety. Also, these three aspects were the main measurements of the pre-test and post-test.

The specific process of this study was to first recruit subjects through WeChat and then screen them according to the UCS criteria set in this study. After screening, 90 university students with UCS were selected for random grouping. This experiment by different intervention methods can be divided into two experimental groups, Baduanjin group and PNF group, and a control group, that is, no intervention group. After the grouping, a pretest was administered to evaluate mainly from neck range of motion, static posture and self-perception. After the pre-test, each group received the experimental intervention treatment for 12 weeks. 12 weeks later a post-test was administered, which was consistent with the pre-test. The final data collected.

ELIGIBILITY:
Inclusion Criteria:

* (1) FHA≥42°; (2) FSA≥49°; (3) Recurrent neck pain accompanied by dizziness and headache for ≥2 months; (4) Chest tightness, easy to panic, dyspnea. Severe cases with dizziness and headache; (5) The neck head is too long at the desk or the pain is aggravated after fatigue; (6) Tenderness and/or spasms in the neck and shoulder; (7) Neck and back muscles are tense and stiff, and neck motion is limited.

Exclusion Criteria:

* (1) Meet the above diagnostic criteria; (2) University students aged 18-23, male or female; (3) No other treatment and no other physical activities during the treatment; (4) Able to complete the whole rehabilitation program as planned; (5) Sign informed consent.

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Static posture | 12 weeks
  Static postures are divided into Forward Head Angle and Forward Shoulder Angle.
Cervical range of motion (CROM) | 12 weeks
  Head forward, head back, head left, head right, head left rotation and head right rotation.
Pain | 12 weeks
  Numeric Pain Rating Scale (NPRS)
Neck disorder | 12 weeks
  Neck Disability Index
Anxiety | 12 weeks
  Self-rating Anxiety Scale
Quality of life | 12 weeks
  SF-12 scale

CONTACTS AND LOCATIONS:
Locations (1):
- Zhengzhou Normal University, Zhengzhou, Henan, China